CLINICAL TRIAL: NCT06075173
Title: PRospEctive Evaluation of DIagnostiC Performances of resTing Full-cycle rAtio in Coronary Bifurcation LEsion (PREDICTABLE Study)
Brief Title: Resting Full-cycle Ratio in Side Branch
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sejong General Hospital (Other)
Collaborators: Soon Chun Hyang University (Other); Keimyung University Dongsan Medical Center (Other); Hanyang University Seoul Hospital (Other)
Responsible Party: Principal Investigator, Hyun Jong Lee, MD, PhD, Sejong General Hospital
Other Study IDs: PREDICTABLE Version 3.5
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Coronary Artery Disease
Keywords: bifurcation lesion; physiologic assessment
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Resting full-cycle ration (RFR) measurments — RFR and FFR measurements in main vessel and side branch lesions
  Other Names: fractional flow ratio (FFR) measurments

SUMMARY:
The goal of this observational study is to evaluate diagnostic performance of resting full-cycle rate (RFR) in side branch lesion.

We aims to evaluate whether the diagnostic performance of RFR in the side branch lesion is non-inferior compared to that in the main vessel lesion RFR and FFR measurements will be performed to define functional significance in patients with side branch lesion with or without main vessel lesion

DETAILED DESCRIPTION:
The presence of myocardial ischemia is the most important prognostic indicator in patients with coronary artery disease. Pressure-based functional assessment has been recommended to assess the presence of myocardial ischemia due to low accuracy of image-based assessment in intermediate coronary artery disease. Selective revascularization for only ischemia-producing lesion with fractinal flow reserve(FFR) guidance proved to decrease adverse cardiac events and avoid unnecessary coronary stenting, compared to angiography-guided revascularization. Therefore, Current guidelines strongly recommend FFR measurement for the assessment of the functional severity of moderate stenosis of a culprit lesion in stable coronary artery disease, and non-culprit lesion in acute coronary syndrome. However, it's clinical adaption in a real world was still very low, because of the need of pressure wire and hyperemic agent. Instantaneous flow ratio (iFR), which the ratio of distal coronary artery pressure to aortic pressure during wave-free period at rest, had a high diagnostic accuracy to define functional significance without need of adenosine. According to two large randomized trials, iFR-guided coronary revascularization proved to be non-inferior to FFR-guided revascularization with respect to one-year risk of major adverse cardiac events. Recently, new adenosine-free index, called as a resting full-cycle ratio (RFR), which is completely independent of the ECG and irrespective of systole or diastole has been validated to detect myocardial ischemia. RFR is not limited by sensitive land marking of components of the pressure waveform unlike iFR, and is diagnostically equivalent to iFR.

This novel physiologic index without need of adenosine have a potential to widely spread of functional assessment for coronary artery stenosis in daily clinical practice, and simplify procedure in complex coronary artery disease. Therefore, we sought to investigate diagnostic performance of this novel physiologic index to define myocardial ischemia in coronary bifurcation lesion, which is one of complex lesion subset.

ELIGIBILITY:
Inclusion Criteria:

* Patients with side branch lesion, who need functional evaluation

Exclusion Criteria:

* Severe LV systolic dysfunction (LVEF <30%)
* Culprit vessel in acute coronary syndrome
* Donor vessel to supply chronic total occlusion lesion of non-target vessel
* Symptomatic valvular heart disease or cardiomyopathy
* Too much overlapping or severe tortuosity to disrupt quantitative coronary analysis
* Previous bypass surgery

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with side branch lesion, who need functional evaluation
Sampling Method: Non-Probability Sample
Enrollment: 286 (Estimated)
Dates: Start 2020-01-08 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
diagnostic sensitivity of RFR in side branch lesions | during index coronary angiography
  diagnostic sensitivity of RFR to predict FFR < 0.80

SECONDARY OUTCOMES:
Specificity, positive predictability, negative predictability, diagnostic accuracy, area under the curve (AUC) value in side branch | during index coronary angiography
  diagnostic performances of RFR to predict FFR < 0.80

CONTACTS AND LOCATIONS:
Locations (1):
- Sejong General Hospital, Bucheon-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No